CLINICAL TRIAL: NCT04156711
Title: Remote Ischemic Preconditioning in Patients Undergoing Acute Minor Abdominal Surgery: The PUMAS Study
Brief Title: Remote Ischemic Preconditioning in Patients Undergoing Acute Minor Abdominal Surgery
Acronym: PUMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REG-020-2019
Record Dates: First submitted 2019-09-23; First posted 2019-11-07 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Acute Cholecystitis; Endothelial Dysfunction
Keywords: Remote ISchemic Preconditioning (RIPC); Acute surgery; Acute cholecystitis; Endothelial dysfunction; Heart Rate Variability (HRV)
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Outcomes assessor are partly blinded and data analysis will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Preconditioning (Experimental): Remote ischemic preconditioning is carried out before the induction of general anesthesia. All four cycles will be completed before general anesthesia. The blood pressure cuff is placed on the upper limb. The cuff is inflated to 200 mmHg (if systolic blood pressures exceeds 185 mmHg, the cuff will be inflated to at least 15 mmHg above the systolic blood pressure) resulting in a total occlusion of the blood flow to the limb. After 5 minutes of ischemia, the cuff is deflated, and the limb is reperfused for 5 minutes. This cycle is repeated 4 times. Pulse oximetry is performed on the RIPC limb to make sure that the blood flow is completely interrupted during ischemia
  Interventions: Procedure: Remote Ischemic Preconditioning (RIPC)
- Control (No Intervention): Will receive no intervention, but will go through same tests at the same time-points (endothelial function measured by reactive hyperemia index, blood samples, Heart rate variability and questionaires)

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning (RIPC) — Cycles of forearm ischemia and reperfusion by the inflation of a blood-pressure cuff over the systemic blood pressure for brief periods
  Arms: Remote Ischemic Preconditioning

SUMMARY:
This study examines if remote ischemic preconditioning in patients undergoing minor acute abdominal surgery (laparoscopic cholecystitis due to acute cholecystitis) is associated with a modulation of endothelial dysfunction. half of the patients will receive remote ischemic preconditioning prior to surgery, the other half will serve as controls.

DETAILED DESCRIPTION:
Remote ischemic preconditioning (RIPC) consists of cycles of forearm or leg ischemia and reperfusion by the inflation of a blood-pressure cuff over the systemic blood pressure for brief periods. The procedure is simple, safe and with no clear side effects. In clinical studies covering acute cardiology RIPC has effectively reduced myocardial injury, postoperative cardiovascular complications and cardiac mortality. Recently, the effect of RIPC on attenuating ischemia-reperfusion injury has been investigated in non-cardiac surgery as well. The organ specific ischemia-reperfusion injury, systemic oxidative stress and inflammatory response were attenuated due to the intervention but a complete understanding of the underlying protective mechanisms of RIPC is however still lacking.

Experimental and clinical studies have implicated that the stimulus of RIPC is transmitted from the preconditioned tissue to other tissues and organs by humoral, neural and systemic anti-inflammatory mediators. The humoral and neural pathway are thought to be dependent on endogen substances such as adenosine, bradykinin, nitrogen oxide (NO) and calcitonin-gene-related-peptide (CGRP).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing acute or subacute cholecystectomy due to acute cholecystitis with a maximum of 7 days of symptoms prior to surgery

Exclusion Criteria:

* Not capable of giving informed consent after oral and written information
* Surgery within 30 days of study inclusion
* Conditions that prevent the performance of remote ischemic preconditioning on the upper extremity, e.g. fractures, paresis, lymphedema
* performance of concomitant endoscopic retrograde cholangiopancreatography (ERCP) during surgery
* synchronous pancreatitis
* synchronous cholangitis

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Changes in endothelial function measured by reactive hyperemia index (RHI) | 24 hours
  Changes in endothelial function measured by reactive hyperemia index (RHI) at baseline, four hours and 24 hours after surgery (cholecystectomy due to acute cholecystitis)

SECONDARY OUTCOMES:
Heart rate variability | 24 hours
  Changes in Heart rate variability measured with eMotion Faros from baseline and 24 hours consecutively.
Changes in p-L-arginine | 24 hours
  Changes in p-L-arginine in μmol/L from baseline til 24h post-surgery
Changes in p-asymmetric dimethylarginine | 24 hours
  Changes in p-asymmetric dimethylarginine in μmol/L from baseline til 24h post-surgery
Changes in p-biopterins | 24 hours
  Changes in p-biopterins in ng/ml from baseline til 24h post-surgery
Changes in soluble endothelial (E-) selectin | 24 hours
  Changes in soluble E-selectin in ng/ml from baseline til 24h post-surgery
Changes in soluble plasma (P-) selectin | 24 hours
  Changes in soluble P-selectin in ng/ml from baseline til 24h post-surgery
Changes in Intercellular Adhesion Molecule 1 (ICAM-1) | 24 hours
  Changes in soluble Intercellular Adhesion Molecule 1 (ICAM-1) in ng/ml from baseline til 24h post-surgery
Changes in syndecan-1 | 24 hours
  Changes in syndecan-1 in pg/ml from baseline til 24h post-surgery
Changes in thrombomodulin | 24 hours
  Changes in thrombomodulin in pg/ml from baseline til 24h post-surgery
Changes in arginine vasopressin | 24 hours
  Changes in arginine vasopressin in ng/ml from baseline til 24h post-surgery
Changes in adrenalin | 24 hours
  Changes in adrenalin in ng/ml from baseline til 24h post-surgery
Changes in noradrenalin | 24 hours
  Changes in noradrenalin in pg/ml from baseline til 24h post-surgery
Changes in ascorbic acid | 24 hours
  Changes in ascorbic acid in ng/μL from baseline til 24h post-surgery
Changes in dehydroascorbic acid | 24 hours
  Changes in dehydroascorbic acid in ng/μL from baseline til 24h post-surgery
Changes in angiotensin II | 24 hours
  Changes in angiotensin II in pg/mL from baseline til 24h post-surgery
Changes in bradykinin | 24 hours
  Changes in bradykinin in pg/mL from baseline til 24h post-surgery
Changes in calcitonin-gene related peptide | 24 hours
  Changes in calcitonin-gene related peptide in pg/mL from baseline til 24h post-surgery
Changes in prostacyclin | 24 hours
  Changes in prostacyclin in pg/mL from baseline til 24h post-surgery
Changes in serotonin | 24 hours
  Changes in serotonin in ng/mL from baseline til 24h post-surgery
Changes in endothelin-1 | 24 hours
  Changes in endothelin-1 in pg/mL from baseline til 24h post-surgery
Changes in adrenomedullin | 24 hours
  Changes in adrenomedullin in ng/mL from baseline til 24h post-surgery
Changes in platelets | 24 hours
  Changes in platelets x 109/L from baseline til 24h post-surgery
Changes in adenosin | 24 hours
  Changes in adenosin μmol/L from baseline til 24h post-surgery
Changes in interleukin-6(IL-6), interleukin-10 (IL-10), tumor necrosis factor alpha (TNF-alpha), transforming growth factor beta (TGF-beta) | 24 hours
  Changes in IL-6, IL-10, TNF-Alpha, TGF-beta in pg/mL from baseline til 24h post-surgery
Changes in gene expression autoimmune human pathway panel from NanoString | 4 hours
  Changes in gene expression profiles in the autoimmune human pathway panel from NanoString from baseline until four hours post-surgery.
Local complications to RIPC | 24 hours
  Pain, changed sensibility or decreased function of the upper extremity where remote ischemic preconditioning were carried out preoperatively.
Differences in postoperative quality of recovery score 15 (QoR-15) between arms in the trial | 30 days
  Questionnaire on Postoperative quality of recovery with 15 questions comparing scores from baseline, 24 hours and 30 days after surgery between study arms (intervention and controls)
Differences in Self reported pain on a 0-10 scale between arms in the trial | 24 hours
  Self reported pain on a 0-10 scale at baseline and 24 hours after surgery between study arms (intervention and controls)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten L Wahlstroem, MD, Principal Investigator — Center for Surgical Science, Zealand University Hospital,
Locations (1):
- Center for Surgical Science, Surgical Department, Zealand University Hospital, Køge, Region Sjælland, Denmark